CLINICAL TRIAL: NCT04068116
Title: Impact of Ischemic Post-conditioning During Primary Percutaneous Coronary Intervention on Left Ventricular Remodeling and Global Systolic Function in Patients Presenting With ST-Elevation Myocardial Infarction
Brief Title: Impact of Ischemic Post-conditioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Fathi Ahmad, Cardiologist, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: ST Elevation Myocardial Infarction; Ventricular Remodeling; Ventricular Dysfunction; Ischemic Reperfusion Injury
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling; Ventricular Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postconditioning in primary percutaneous coronary intervention (Experimental): Patients presenting with ST-elevation myocardial infarction will undergo primary per-cutaneous coronary intervention with post-conditioning by making 4 cycles of repeated occlusion & re-perfusion 30-second each by inflation/deflation of an appropriately sized PTCA (per-cutaneous trans-luminal coronary angioplasty) balloon
  Interventions: Procedure: Primary per-cutaneous coronary intervention
- Primary percutaneous coronary intervention (Active Comparator): Patients presenting with ST-elevation myocardial infarction will undergo primary per-cutaneous coronary intervention without post-conditioning
  Interventions: Procedure: Primary per-cutaneous coronary intervention

INTERVENTIONS:
Procedure: Primary per-cutaneous coronary intervention — Patients presenting with ST-elevation myocardial infarction will undergo primary per-cutaneous coronary intervention including balloon angioplasty & coronary stent deployment as needed +/- post-conditioning (for post-conditioning arm) making 4 cycles of repeated occlusion & reperfusion 30-second each by inflation/deflation of an appropriately sized PTCA (percutaneous transluminal coronary angioplasty) balloon

SUMMARY:
Study will investigate & compare the left ventricular remodeling & systolic function between two groups of ST-elevation myocardial infarction undergoing primary per-cutaneous coronary intervention applying ischemic post-conditioning to one of them.

DETAILED DESCRIPTION:
Among re-perfusion strategies for the management of ST-elevation myocardial infarction , primary per-cutaneous coronary intervention is the preferred one within 120 minutes from the first medical contact.However , restoration of the coronary blood flow can paradoxically reduce the beneficial effects of myocardial re-perfusion , a phenomenon known as myocardial re-perfusion injury.Ischemic post-conditioning has been described as a measure for myocardial salvage , performed by making cycles of briefly interrupted perfusion during the early moments of coronary re-flow.Post-conditioning may be performed immediately after the early re-flow by creating cycles of interrupted inflation & deflation of the angioplasty balloon in patients undergoing primary per-cutaneous coronary intervention.In this study investigators aim to compare the left ventricular remodeling and global systolic function immediately & 6 months after re-perfusion between two groups of 100 patients presenting with acute ST-elevation myocardial infarction, using ischemic post-conditioning in one group of patients undergoing primary per-cutaneous coronary intervention (n=50 patients) by making 4 cycles of repeated occlusion & re-perfusion 30-second each by inflation/deflation of an appropriately sized per-cutaneous trans-luminal coronary angioplasty balloon.The other group will be investigated after re-perfusion by primary per-cutaneous coronary intervention without ischemic post-conditioning (n=50 patients)

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with symptoms of acute myocardial ischemia with time of symptom onset < 12 hours & meeting the other following criteria of type 1 myocardial infarction according to the fouth universal definition of myocardial infarction(Thygesen, 2019):

   * Detection of a rise and/or fall of cardiac troponin values with at least one value above the 99th percentile upper reference limit.(URL)
   * Ischemic ECG changes; New or persistent ST-segment elevation with development of pathological Q waves
   * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic etiology.
2. Patients undergoing primary percutaneous coronary intervention as the first choice of revascularization therapy.

Exclusion Criteria:

1. Patients with transient ST segment elevation in the surface electrocardiography.
2. Patients presenting within > 12 hours from the onset of maximal symptoms.
3. Patients with evidence of pre-infarction angina.
4. Patients with evidence of collateral blood flow to the infarct region on their angiogram.
5. Patients with history of old myocardial infarction causing chronic impairment of LV systolic function.
6. Patients presenting with ST-segment elevation myocardial infarction other than type 1 according to the fouth universal definition of myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Left ventricular remodeling | Immediate-6 months
  percentage of increase in left ventricular end-diastolic volume (EDV) and/or left ventricular end-systolic volume (ESV)

OTHER OUTCOMES:
Left ventricular Ejection Fraction | Immediate-6 months
  is a simple measure of global systolic function that pervades the risk evaluation and management of many cardiovascular diseases